CLINICAL TRIAL: NCT05578300
Title: Effective Translation of Endovascular Thrombectomy Trials Into Real-world Practice in the Asia-Pacific: a Multicenter, Prospective Registry (ENDURE-APAC)
Brief Title: Effective Translation of Endovascular Thrombectomy Trials Into Real-world Practice in the Asia-Pacific
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Linyi People's Hospital (Other)
Responsible Party: Principal Investigator, Dr. IP Yiu Ming Bonaventure, Assistant Professor, Chinese University of Hong Kong
Other Study IDs: CREC 2022.414
Record Dates: First submitted 2022-10-11; First posted 2022-10-13 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Ischemic Stroke; Stroke; Stroke, Acute; Stroke, Ischemic; Brain Diseases; Major Adverse Cardiovascular Event
MeSH Terms: conditions — Ischemic Stroke; Stroke; Brain Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Physical, histology, biochemical or protein expressions of the thrombi obtained from thrombectomy procedures may contain information regarding the etiology of stroke and relevant disease pathology. The investigators shall store the thrombus, if any, yielded from thrombectomy procedures for future analyses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with ischemic stroke with suspected large vessel occlusion: The investigators shall recruit patients that meet the following inclusion criteria:
  1. Patient who are over 18 years of age.
  2. Patient with ischemic stroke with suspected large vessel occlusion (LVO), defined as occlusion of the internal carotid artery (ICA), M1 or M2 segment of the middle cerebral artery (MCA), or basilar artery (BA).
  Interventions: Diagnostic Test: Thrombus analyses; Diagnostic Test: Imaging assessment

INTERVENTIONS:
Diagnostic Test: Thrombus analyses — Physical, histology, biochemical or protein expressions of the thrombi obtained from thrombectomy procedures may contain information regarding the etiology of stroke and relevant disease pathology. The investigators shall store the thrombus, if any, yielded from thrombectomy procedures for future analyses.
Diagnostic Test: Imaging assessment — All imaging data will be deidentified before assessment. Plain computer tomography of the brain (CT brain), CT angiography (CTA), CT perfusion (CTP), magnetic resonance imaging of the brain (MRI), digital subtraction imaging (DSA) will be analysed. The investigators shall blind the assessors from treatment choice and outcome in all analyses that require human assessment.

SUMMARY:
As a major breakthrough of acute stroke treatment over the past decade, endovascular thrombectomy (EVT) drastically improved neurological recovery and survival in patients with large vessel occlusion (LVO) ischemic strokes in major clinical trials. Nevertheless, much remained uncertain about the implementation of scientific evidence of EVT into real-world benefits. For instance, healthcare policies that influence critical time-matrices, endovascular thrombectomy techniques that may enhance success rate or prevent complications, or advanced imaging techniques that allow precise prognosis or expansion of treatment populations, should be evaluated. On the other hand, capturing LVO patients who were not able to undergo EVT may reveal the gap between clinical trials and real-world practice in the Asia-Pacific.

In this multicenter prospective collaboration across the Asian-Pacific, the investigators aim to evaluate the determinants of effective EVT in the real-world setting.

DETAILED DESCRIPTION:
In this multicenter, prospective, longitudinal study, the investigators aim to evaluate the determinants of effective EVT in the real-world setting.

The investigators shall recruit patient who are over 18 years of age, with ischemic stroke with suspected large vessel occlusion (LVO), defined as occlusion of the internal carotid artery (ICA), M1 or M2 segment of the middle cerebral artery (MCA), or basilar artery (BA).

Detailed study procedures are as follows:

1. As the EVT center of the New Territory East Cluster (NTEC), all patients who undergo EVT triage in the NTEC, i.e. patients with suspected LVO, would be assessed by neuro-interventionists from the Prince of Wales Hospital (PWH). Eligibility screening for recruitment under the ENDURE-APAC registry will be carried out simultaneously.
2. The investigators shall obtain informed consent either from patient or next-of-kin. Informed consent will be obtained from his/her legal guardian or next-of-kin for those incompetent subjects who are willing to participate in the study. Subjects will be reconsented when competent.
3. After the informed consent, a study identity number will be assigned to each participant. The investigators shall obtain the following data:

   1. Demographic data such as age, gender, date of birth, smoking and drinking habit, pre-morbid functional status (by modified Rankin Scale (mRS)).
   2. Co-morbidities including hypertension, diabetes mellitus, hyperlipidemia, atrial fibrillation, previous strokes, ischemic heart disease, peripheral vascular disease, congestive heart failure, etc.
   3. Concurrent medications including anticoagulants (apixaban, dabigatran, edoxaban, rivaroxaban, heparin, warfarin), antiplatelet agents (aspirin, clopidogrel, ticagrelor, cilostazol), lipid-lowering agents (simvastatin, atorvastatin, rosuvastatin, pravastatin, fluvastatin, ezetimibe, gemfibrozil, fenofibrate, erenumab), antihypertensive (angiotensin converting enzyme inhibitors, angiotensin receptor blockers, beta blockers, calcium channel blockers, diuretics, aldosterone antagonists, nitrates, etc.), cytochrome P450 or P-glycoprotein inhibitors (amiodarone, dronedarone, phenytoin, valproate, carbamazepine, levetiracetam, rifampicin, cyclosporin, etc.), non-steroidal anti-inflammatory agents or cyclo-oxygenase2 inhibitors (indomethacin, ibuprofen, diclofenac, celecoxib, etorixocib), glucose lowering drugs (metformin, gliclazide, glimepiride, empagliflozin, dapagliflozin, insulin, exenatide, semaglutide, liraglutide, dulaglutide).
   4. Radiological findings, treatment outcomes and complications (see 2.3.2 and 2.3.4.) will be documented.
   5. Baseline hemoglobin, white blood cell, platelet count, creatinine, sodium, potassium, alanine transferase, alkaline phosphatase, high density lipoprotein cholesterol, low density lipoprotein cholesterol, total cholesterol, triglyceride level, prothrombin time, activated thromboplastin time, fasting glucose, glycated hemoglobin A1c will be documented.

ELIGIBILITY:
Inclusion Criteria:

* Patient who are over 18 years of age.
* Patient with ischemic stroke with suspected large vessel occlusion (LVO), defined as occlusion of the internal carotid artery (ICA), M1 or M2 segment of the middle cerebral artery (MCA), or basilar artery (BA).

Exclusion Criteria:

* Patient with isolated vertebral artery occlusion not involving the BA.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese Stroke Population
Sampling Method: Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2022-10-21 (Actual); Primary Completion 2032-10-20 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Pre-morbid functional status assessed by modified Rankin Scale (mRS) | 18 October 2032
  Neurological recover and survival as assessed by mRS at 90 days, with the scale runs from 0-6, running from perfect health without symptoms (Score 0) to death (Score 6).

CONTACTS AND LOCATIONS:
Overall Officials: Bonaventure Yiu Ming IP, MB ChB, Principal Investigator — Chinese University of Hong Kong
Locations (3):
- China (2):
  - Linyi People's Hospital, Linyi, Shandong
  - The Affiliated Hospital of Medical College of Qingdao University, Qingdao, Shandong
- Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No